CLINICAL TRIAL: NCT03594461
Title: Intense Treatment Regimen With Intravitreal Aflibercept Injection for Refractory Neovascular Age-Related Macular Degeneration With or Without Polypoidal Choroidal Vasculopathy
Brief Title: Intense Treatment Regimen With Intravitreal Aflibercept Injection
Acronym: I-TRAP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-TRAP
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2mg IAI q2w (Experimental): 2mg Intravitreal Aflibercept injection will be given every 2 weeks starting at baseline and then at weeks 2, 4, 6, 8, 10 and 12. Patients will then be seen at week 16 (4 weeks following the end of the intensive dosing period), and a treat and extend regimen will be initiated through week 52.
  Interventions: Drug: Aflibercept Injection
- 2mg IAI q3w (Experimental): 2mg Intravitreal Aflibercept injection will be given every 3 weeks starting at baseline and then at weeks 3, 6, 9 and 12. Patients will then be seen at week 16 (4 weeks following the end of the intensive dosing period), and a treat and extend regimen will be initiated through week 52.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Intense Treatment Regimen for Refractory Neovascular Age-Related Macular Degeneration with or without Polypoidal Choroidal Vasculopathy
  Other Names: Eylea

SUMMARY:
This study will evaluate the safety and efficacy of intense dosing for a limited period in patients who demonstrate refractory disease on monthly IAI. Patients will be followed for 52 weeks

DETAILED DESCRIPTION:
The development of biologic therapy targeting VEGF has been revolutionary and has lowered the rate of functional blindness in many developed countries. Modalities to treat nvAMD have been based on monthly dosing. For many patients, this modality is adequate and they can achieve a dry macula. A subset of patients can even have their treatment intervals extended. There is, however, a subset of patients with recalcitrant neovascularization for whom IAI fails to produce a dry macula even with q4w dosing. An intense dosing schedule for a short period of time could decrease fluid activity in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Choroidal neovascularization related to age-related macular degeneration
* Prior treatment with any anti-VEGF agent for ≥ 12 months
* Prior treatment with at least five consecutive IAI at baseline with an average treatment interval of maximum 35 days
* Presence of foveal fluid at most recent clinical visit occurring 30 (+/- 5) days following the most recent IAI
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

* Monocular patients
* Patients with a previous history of macular thermal laser or PDT
* Confounding ocular conditions in the study eye that may affect interpretation of OCT, BCVA or assessment of macular appearance (eg. cataract, epiretinal membrane, retinal vascular occlusive disease)
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding baseline
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Active intraocular inflammation (grade trace or above) in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment
* Patients on systemic anti-VEGF treatment
* Pregnant or breastfeeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception prior to the initial dose/start of the first treatment, during the study, and for at least 3 months after the last dose. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly.

  * *Contraception is not required for men with documented vasectomy.
  * **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and non ocular adverse events through to week 12 of intensive IAI therapy | Baseline to 12 weeks

SECONDARY OUTCOMES:
Mean change in BCVA from baseline to week 12 | Baseline to week 12
Mean change in BCVA from baseline to week 52 | Baseline to week 52
Number of patients who are able to maintain a dry macula with IAI intervals extending beyond q4w. | Baseline to week 52
Mean number of injections to achieve fluid-free status and at week 12 and week 52 | Baseline to week 52
Incidence and severity of adverse events through week 52 | Baseline to week 52
Polyp size reduction or closure - compare polyp and lesion area size to baseline on Heidelberg Eye Explorer software (Tan 2015), OCTA and ICG angiography (ICGA) | Baseline to week 52
Mean change to area of flow within neovascular network on OCT-angiography (OCTA) | Baseline to week 12
Mean change to area of flow within neovascular network on OCT-angiography (OCTA) | Baseline to week 52
Mean change in lesion | Baseline to week 12
Mean change in lesion | Baseline to week 52
Number of patients whose fovea remain dry upon extending to q4w IAI at week 52 | Baseline to week 52
Number of patients whose subfoveal fluid is resolved or with no further increase in extrafoveal fluid | Baseline to week 12
Number of patients whose subfoveal fluid is resolved or with no further increase in extrafoveal fluid | Baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: K. Bailey Freund, MD, Principal Investigator — Vitreous -Retina- Macula Consultants of New York
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided